CLINICAL TRIAL: NCT01677234
Title: Comparison of Arm and Forearm Blood Pressure During Elective Cesarean Delivery
Brief Title: Wrist NIBP During Elective Cesarean Delivery
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: H12-01797
Record Dates: First submitted 2012-08-29; First posted 2012-08-31 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: Wrist Blood Pressure Measurements; Anesthesia Resulting in Shivering
Keywords: Blood pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant women: Pregnant women undergoing a cesarean section

SUMMARY:
Blood pressure is typically measured with a non-invasive cuff placed on the upper arm. This cuff cannot take accurate measurements when the patient's arm is moving. Anesthesia for a cesarean delivery frequently causes the patient to shiver and their arm to shake, and sometimes to the extent that blood pressure cannot be measured. A cuff placed on the wrist may be more effective when a patient is shivering because their lower arm moves less and can be more easily stabilized. We will be taking simultaneous blood pressure measurements both just before and during cesarean deliveries in order to compare blood pressure at the upper arm versus the wrist.

DETAILED DESCRIPTION:
Upper arm non-invasive blood pressure (NIBP) measurement is the most commonly accepted method of blood pressure (BP) monitoring. During a cesarean delivery it may be challenging to obtain an accurate measurement from the automated devices in over 50% of the attempts due to arm movement.1 Patients may voluntarily move their arm, but more often neuraxial (spinal, epidural, combined spinal-epidural) anesthesia is known to induce shivering that causes the patient's arm to shake.2 To eliminate the effect of movement of the upper arm, NIBP has been tested on the leg because it is immobilized during neuraxial anesthesia. However, studies monitoring NIBP on an ankle or a calf were unable to accurately detect changes (increase or decrease) in blood pressure in patients undergoing a cesarean delivery.3,4 It seems clinically reasonable that in the case of a shivering patient, the forearm, with less muscle mass, would shake less and could be stabilized more easily than the upper arm (stabilizing the forearm is easily done by holding the patient's hand with a light pressure on the arm rest). Therefore, positioning an NIBP cuff on the forearm (near the wrist) may be useful to obtain an accurate blood pressure measurement in shivering patients.

Previous studies have found that forearm BP overestimates blood pressure measured at the upper arm in a variety of clinical settings and patient populations under static (patient at rest, not submitted to an intervention that might alter BP) circumstances.5-8 It is unknown whether this overestimation is clinically relevant when blood pressure change occurs rapidly, such as during a cesarean delivery. During neuraxial anesthesia for cesarean delivery, it is important for the anesthesiologist to know both absolute values and clinically significant changes in blood pressure to determine their treatment. The detection of dynamic changes in blood pressure (as when the patient is submitted to an intervention that might alter BP per se, e.g. neuraxial anesthesia) has been studied in obstetric patients. Nevertheless, either due to the location where the BP cuff was placed4 (as on the lower limb with interference of the aorto-caval compression) or to the technology used to measure blood pressure,9 (the penaz technology was not consistent with oscillometric technology in a previous study) the forearm blood pressure was not comparable to upper arm blood pressure when measured using an oscillometric monitor.

This study will compare the upper arm (the current gold-standard) and the forearm NIBP measurements in patients undergoing an elective cesarean delivery under subarachnoid anesthesia. We hypothesize that the forearm systolic BP measurement values will be within 10% (lower or higher) of the systolic BP values measured in the upper arm at the same time-points

ELIGIBILITY:
Inclusion Criteria:

* Healthy (American Society of Anesthesiologist's (ASA) physical status I or II) patients
* Having an elective cesarean delivery under spinal or combined spinal epidural anesthesia
* ≥19 years old

Exclusion Criteria:

* Contra-indication to neuraxial anesthesia
* General anesthesia for any reason prior to delivery of the baby
* Use of the epidural component (epidural top-up) of combined spinal epidural anesthesia (prior to delivery of the baby)
* History of cardiovascular disease, e.g. hypertension (either essential or pregnancy-induced)
* A difference of more than 10% between both upper arms and forearms in mean blood pressure measurement prior to surgery (see below)
* BMI >35kg/m2 (it is more difficult to ensure the cuff size is correct in these obese patients)
* Inability to read and understand English for the purpose of informed consent

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women having an elective cesarean delivery at BC Women's Hospital in Vancouver, British Columbia.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2012-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Compare trends in NIBP measurements between the upper arm and forearm | 30 minutes
  Measure NIBP at the upper arm and forearm simultaneously during surgery. NIBP cuffs will be on opposite arms.

SECONDARY OUTCOMES:
To estimate the accuracy of blood pressure measured on the forearm | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Simon Massey, MD, Principal Investigator — University of British Columbia, BC Women's Hospital
Locations (1):
- British Columbia's Women's Hospital, Vancouver, British Columbia, Canada